CLINICAL TRIAL: NCT04406285
Title: Effects of Periodized and Autoregulated Resistance Training Programs in Haematological Cancer Patients Undergoing High-dose Chemotherapy and Hematopoietic Stem Cell Transplantation: A Randomized, Controlled Clinical Trial.
Brief Title: Effects of Periodized and Autoregulated Resistance Training in Haematological Cancer Patients During the Treatent.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Fabrício Edler Macagnan, Sponsor-Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TMO-2019
Record Dates: First submitted 2020-05-14; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Fatigue; Leukemia; Lymphoma; Physical Disability
Keywords: Fatigue; Physical Therapy; Hematological Malignancy
MeSH Terms: conditions — Fatigue; Leukemia; Lymphoma; Hematologic Neoplasms | interventions — AIEOP acute lymphoblastic leukemia protocol

STUDY DESIGN:
Intervention Model Description: Patients will be included sequentially by convenience (according to the inclusion and exclusion criteria) in non-probabilistic form. The included individuals will be randomized by Random Allocation System software in two separate lists: one for patients diagnosed with leukemia (subdivided into a control and experimental group) and other for patients diagnosed with lymphoma (equally divided into a control and experimental group). The allocation ratio will be 1/1 in order to maintain balance in division between control and experimental groups. On the other hand, balancing the different clinical diagnoses will depend on chance, even though the historical average of the service shows similar proportions in the number of cases treated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Leukemia Control Group (Active Comparator): In this group the exercise program will be based on the standard protocol of physical therapy.
  Interventions: Other: Standard protocol Leukemia
- Leukemia Experimental Group (Experimental): In this group the exercise program will be based on a periodic resistance training program, with an autoregulated approach within a non-linear model, based on the individual's patient daily response.
  Interventions: Other: Periodic Resistance Training Program Leukemia
- Lymphoma Control Group (Active Comparator): In this group the exercise program will be based on the standard protocol of physical therapy.
  Interventions: Other: Standard protocol Lymphoma
- Lymphoma Experimental Group (Experimental): In this group the exercise program will be based on a periodic resistance training program, with an autoregulated approach within a non-linear model, based on the individual's patient daily response.
  Interventions: Other: Periodic Resistance Training Program Lymphoma

INTERVENTIONS:
Other: Standard protocol Leukemia — * Bicycle ergometer endurance training for 5 minutes, with resistance individually adjusted based on the patient´s feedback (from 70% of maximum heart rate);
  * Resistance exercises for muscle groups: hip flexors, knee extensors and ankle plantar flexors (10 repetitions, 1 sets);
  * Resistance training for arms, using 0,5 kg or 1,0 kg dumbbels (10 repetitions, 1 sets).
  Arms: Leukemia Control Group
Other: Periodic Resistance Training Program Leukemia — * Submaximal Ergometer tests with incremental load (from 85% of maximum heart rate or maximum effort related);
  * 30-Second Chair Stand;
  * Hand Grip Strength and submaximal arm effort using 0,5 kg or 1,0 kg dumbbels.
  Arms: Leukemia Experimental Group
Other: Standard protocol Lymphoma — * Bicycle ergometer endurance training for 5 minutes, with resistance individually adjusted based on the patient´s feedback (from 70% of maximum heart rate);
  * Resistance exercises for muscle groups: hip flexors, knee extensors and ankle plantar flexors (10 repetitions, 1 sets);
  * Resistance training for arms, using 0,5 kg or 1,0 kg dumbbels (10 repetitions, 1 sets).
  Arms: Lymphoma Control Group
Other: Periodic Resistance Training Program Lymphoma — * Submaximal Ergometer tests with incremental load (from 85% of maximum heart rate or maximum effort related);
  * 30-Second Chair Stand;
  * Hand Grip Strength and submaximal arm effort using 0,5 kg or 1,0 kg dumbbels.
  Arms: Lymphoma Experimental Group

SUMMARY:
Several clinical trials have demonstrated the positive impact of physical functioning and fatigue in patients who received training programs during the myeloablative chemotherapy with stem cell transplantation. However, the heterogeneity among the forms of physical activity results in moderate to very low evidence available about benefits of physical exercise. In this randomized and controlled clinical trial, we will study the effects on physical performance and fatigue of periodic resistance training programs, with an autoregulated approach within a non-linear model, based on the individual patient response to cancer treatment.

DETAILED DESCRIPTION:
The sample will consist of 66 patients diagnosed with leukemia and lymphoma undergoing high-dose chemotherapy, with or without hematopoietic stem cell transplantation, who will be randomized into two groups. The physical performance and fatigue outcomes will be compared between the control and the experimental group. The control group will perform an exercise program based on the standard protocol of physical therapy, consisting of bicycle ergometer endurance training for 5 minutes, with resistance individually adjusted based on the patient's feedback (from 70% of maximum heart rate) and resistance exercises for muscle groups hip flexors, knee extensors and ankle plantar flexors and resistance training form arms, with weigths of 0,5 to 1,0 kg (10 repetitions, 1 set).

The experimental group will perform a periodic resistance training program, with an auto-regulated and a non-linear model, using the Submaximal Ergometer tests with incremental load (from 85% of maximaum heart rate or maximum effort related), 30-Second Chair Stand, Hand Grip strenght and submaximal effort of arms with weights of 0,5 to 1,0 kg.

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically diagnosed with Leukemia or Lymphoma, in the first or second line of treatment, undergoing high-dose chemotherapy, with or without hematopoietic stem cell transplantation;
* Neurological and cognitive functions preserved;
* Physical conditions that enable participation in physical rehabilitation.

Exclusion Criteria:

* Clinical Complications that contraindicate physical therapy exercises, including the practice of cycle ergometer and resistance exercises;
* Previous musculoskeletal alteration that interferes in physical performance evaluation tests;
* Recent cardiovascular or pulmonary disease;
* Psychiatric or neurological disorder;
* Inability to walk on its own or presence of bone metastasis;
* Adherence on less than 50% of the total sessions of the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Fatigue | Trough study completion, an average of 17 months
  Piper Fatigue Scale, developed by Piper et al. (1998), is a multidimensional measure of fatigue in the field of cancer research and includes subdomains of the behavioral, affective, sensorial and cognitive attributes / fatigue mood, composed of 22 items. The scores for each item range from 0 to 10 and can total 220 points. Higher values characterize a greater perception of fatigue. It will be applied on patient's evaluation day and on hospital discharge day.
Physical Functioning Maximum Capacity | Trough study completion, an average of 17 months
  To evaluate the maximum capacity and endurance of the participants of this study, based on the concept of periodization (volume, intensity and frequency) and self-regulation (volume, intensity and magnitude according to daily readiness of the patient), by Fairman et al., (2017), the patient will perform a submaximal incremental exercise test in a cycle ergometer with electromagnetic braking, keeping the cadence fixed throughout the whole period of the test; the workload will be adjusted progressively every 1 minute until it reaches 85% of maximum heart rate or until the patient reports fatigue. At each load increase, the evaluation of the perceived effort will be performed through the BORG scale. The load, time and distance variables will be evaluated daily.
Lower Limb Physical Functioning and Strength | Trough study completion, an average of 17 months
  The 30-Second Chair Stand evaluates lower limb strength and, indirectly, the risk of falls, especially in the elderly population (JONES, J., RIKLI, 2002). This way, it will compose the set of tests used to determine the physical performance by measuring the number of stands from an armless chair of standard height (45 cm) performed in 30 seconds. The test will be begin when the participant, seating on a neutral spine position and feet flat on the floor, will be instructed to rise to a full stand and return to the original seated position, as quickly as possible. The participant will be instructed to move at maximal speed until they either feel the need to stop or the 30-second time limit is reached. More than 8 unassisted stands for men and women are considered above average for their age, and those below the range as below average.
Handgrip Strength Physical Functioning | Trough study completion, an average of 17 months
  A standard adjustable-handle hydraulic dynamometer will be used to measure hand grip strength as an index of upper limb strength. The Jamar® dynamometer, developed by Bechtol (1954), is considered the most accepted instrument ("gold standard") and is recommended by the American Society of Hand Therapists (ASHT) for being simple, to enable a quick and direct reading of the data and to enable its use in different fields of research. Three measurements of the manual grip strength should be performed in both hands, considering that the maximum difference between them does not exceed 10%, and the average of these being considered as the maximum value.

SECONDARY OUTCOMES:
Healt-related quality of life: EORTC QLQ-C30 | Trough study completion, an average of 17 months
  General health-related quality of life will be assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30), created as an initiative of the Quality of Life Group, from the EORTC (Aaronson et al., 1993) to assess the quality of life of cancer patients. The instrument is composed of 30 items, divided into five functioning scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), one scale that evaluates overall quality of life, five single terms (dyspnea, sleep disturbance, appetite loss, constipation, and diarrhea), and one separate item to evaluate financial impact. Responses are given on a 4-point Likert scale, except for the items that evaluate overall quality of life (items 29 and 30), which are given on a 7-point Likert scale. It will be applied on the day of the patient's evaluation and on the day of hospital discharge.
Symptoms Assessment | Trough study completion, an average of 17 months
  The Edmonton Symptom Assessment Scalemorning will be applied to eavaluate symptoms of pain, tiredness, drowsiness, appetite, nausea, shortness of breath, depression, anxiety and well-being. It is a scale where the patient provides an auto-report on a score that can vary from 0 to 10, being score 0 absence of symptoms and 10 represents the most intense sensation experienced by the patient.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Fabrício Edler Macagnan, Porto Alegre, Rio Grande do Sul
  - Universidade Federal de Ciências da Saúde de Porto Alegre, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No